CLINICAL TRIAL: NCT03735693
Title: Diagnosis of Muscular Weakness Syndrome After a Stay in Intensive Care : Measurement by Ultrasound
Acronym: FIBER
Status: Terminated | Type: Observational
Why Stopped: missing data, little recruitment
Sponsor: Association Pro-arte (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2018-FIBER
Record Dates: First submitted 2018-10-30; First posted 2018-11-08 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-11

CONDITIONS: Amyotrophia; Weakness, Muscle
Keywords: ultrasound; intensive care
MeSH Terms: conditions — Muscular Atrophy; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ulstrasound — measurement of right femoral cross-section

SUMMARY:
The objective is to diagnose earlier and more precisely the occurrence of a weakness neuromuscular syndrome at the end of intensive care, or within 28 days if the stay is longer than 28 days. The amyotrophy has been shown to be proportional to muscle strength in healthy subjects. The amyotrophy can be reliably evaluated by measuring the cross-sectional area of the right femoral muscle. The hypothesis is that amyotrophy measured by muscle ultrasound can allow an early and reliable diagnosis of neuromuscular weakness syndrome (NMWS), even though the measurement of the MRC score (the Gold Standard), has shown its limitations in intensive care in terms of reliability and delayed diagnosis.

Moreover, this syndrome is associated with a loss of functionality and a deterioration of long-term quality of life. One of the objectives is thus to determine if the muscular ultrasound allows a prediction of the occurrence of these alterations far from the intensive care.

Early rehabilitation has shown a benefit on mortality, duration of stay, mechanical ventilation and on functional alteration after intensive care. This is why an earlier and more precise means of diagnostic of this pathology is searched.

The target population is therefore patients from 18 to 80 years hospitalized in intensive care for prolonged stay (> 5 days), and prolonged ventilation (> 48H).

DETAILED DESCRIPTION:
Neuromuscular weakness syndrome post intensive care is a generalized muscular weakness with amyotrophy caused by the stay in the intensive care unit. This pathology is frequent, under diagnosed, increases the length of stay and mortality in intensive care and alters the functional status in the long term (mobility, autonomy, cognitive abilities). The gold standard is the MRC score. It must be under 48/60. But this means of diagnostic is unreliable and tardive (problem of voluntary cooperation, confusion, sedation).

This study allows the earlier diagnosis of neuromuscular weakness syndrome, by muscular ultrasound. Ultrasound of the right femoral muscle allows evaluation of the amyotrophy, which is related to the maximum muscular strength.

The early rehabilitation enable improved prognosis. This is an observational, prospective, single-center, blinded, observational study.

The objective is to determine the day of ultrasound examination with the highest diagnostic performance to predict with a maximum of specificity the occurrence of post-intensive care neuromuscular weakness syndrome, defined by an MRC score <48/60 at the end of intensive care or if the duration of stay exceeds 28 days on the 28th day of hospitalization in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Predictable mechanical ventilation time of at least 48 hours
* Patient intubated for less than 48 hours
* Social security
* Not opposing, or whose family does not object to this research

Exclusion Criteria:

* Neuromuscular pathology
* Amputation of one of the limbs
* Central or peripheral neurological impairment impacting the realization of the MRC score
* Orthopaedic trauma of the limbs or the pelvis preventing the achievement of an MRC score at the exit of resuscitation or by default at J28
* Subject in exclusion period of another study
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns people admitted in intensive care unit, intubated and ventilated.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Determination of the day of ultrasound examination having the highest diagnostic performance to predict with a maximum of specificity the occurrence of a neuromuscular weakness syndrome post-intensive care unit | through study completion, an average of 1 year
  Two-to-two comparison of the AUCs of 3 ROC curves corresponding to 3 measurements by ultrasound of decreasing muscles between J1-J5, J1-J7 and J1-J10

SECONDARY OUTCOMES:
Determination of the perfect threshold of muscular decrease allowing the prediction with the maximum of specificity of a post-intensive care neuromuscular weakness syndrome | through study completion, an average of 1 year
  Look for the 3 ROC curves corresponding to 3 measurements of ultrasound muscle reduction between J1-J5, J1-J7 and J1-J10, the optimal threshold for measuring the cross sectional area of the right femoral muscle
comparison of the persistence of neuromuscular weakness into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | 3 months after discharge from hospital
  MRC score : Medical Research Council (muscular testing), from 0 to 5 for each muscular group, and from 0 (complete tetraplegia) to 60 (normal muscular strength) for the total. The 6 subscales are summed.
comparison of functional alteration into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | 3 months after discharge from hospital
  SF12 score (short form - 12) : quality of life questionnaire, range from 0 to 100. Each standardized data are summed
comparison of functional alteration into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | 3 months after discharge from hospital
  walk test of 6 minuts (Detect abnormalities of gas exchange during exercise)
comparison of functional alteration into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | 3 months after discharge from hospital
  Get up and Go test (evaluates sit-stand transfers, walking, and patient directional changes) : ranges from 1 (no instability) to 5 (very abnormal)
comparison of functional alteration into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | 3 months after discharge from hospital
  ADL score (autonomy scale) : ranging from 0 (dependant) to 6 (independent)
comparison of functional alteration into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | 3 months after discharge from hospital
  the Karnofsky index (description of the general condition of the patient) : from 0% (dead) to 100% (normal state)
comparison of mortality at discharge of intensive care unit into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | during hospitalization in intensive care, at hospital discharge, and 3 months after hospital discharge
  mortality rate
Comparison of length of stay in intensive care unit and hospital into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | through study completion, an average of 1 year
  calculation of the length of stay
Comparison of duration of mechanical ventilation, Optiflow, NIV, and number of days without ventilation into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | through study completion, an average of 1 year
  calculation of the duration of ventilation and no-ventilation
Comparison of malnutrition into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | at intensive care discharge, within a limit of 28 days, at 3 months
  Variation of albuminemia
Comparison of malnutrition into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | at intensive care discharge, within a limit of 28 days, at 3 months
  Variation of pre-albuminemia
Comparison of malnutrition into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | at intensive care discharge, within a limit of 28 days, at 3 months
  Variation of creatinine
Comparison of malnutrition into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | at intensive care discharge, within a limit of 28 days, at 3 months
  Variation of weight
Comparison of malnutrition into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | at intensive care discharge, within a limit of 28 days, at 3 months
  Variation of arm circumference
Comparison of malnutrition into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | at intensive care discharge, within a limit of 28 days, at 3 months
  Variation NUTRIC score ; ranging from 0 (low malnutrition risk) to 10 (the most likely to benefit from aggressive nutrition therapy).
Comparison of calorie intake into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | through study completion, an average of 1 year
  Daily calorie intake
Comparison of drug intake into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | through study completion, an average of 1 year
  the number of days with sedation in intensive care
Comparison of drug intake into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | through study completion, an average of 1 year
  the number of days with curarization in intensive care
Comparison of drug intake into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | through study completion, an average of 1 year
  the dose of opioids in intensive care
Comparison of drug intake into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | During stay in intensive care
  the number of days with sedation and curarization in intensive care, the dose of opioids and the administration of corticosteroids in intensive care
Comparison of drug intake into 2 cohorts of patients (probably not affected by the syndrome, and probably affected) | through study completion, an average of 1 year
  the administration of corticosteroids in intensive care

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available to other researchers